CLINICAL TRIAL: NCT02739659
Title: Carbon Ion Radiotherapy for the Treatment of Localized Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Qing Zhang,MD, DIRECTOR, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-PCa 2015-01
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Prostate Carcinoma
Keywords: prostate carcinoma; carbon-ion radiotherapy; efficacy; toxicity
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Heavy Ion Radiotherapy

ARMS (1):
- carbon-ion radiotherapy (Experimental): Five dose levels [59.2 GyE(Gray equivalent)/16Fx, 60.8 GyE/16Fx, 62.4 GyE/16Fx, 64.0 GyE/16Fx and 65.6 GyE/16Fx] are planned within the Phase I part. After the recommended dose (RD), i.e., MTD, is determined or if the treatments to 65.6 GyE/16Fx are safely delivered, the recommended dose (or 65.6 GyE/16Fx) will be the prescribed dose in the Phase II part of the study.
  Interventions: Device: carbon-ion radiotherapy

INTERVENTIONS:
Device: carbon-ion radiotherapy

SUMMARY:
The aim of this research project is to assess the feasibility and safety of carbon-ion radiotherapy (CIRT) for the treatment of in Chinese localized prostate cancer

DETAILED DESCRIPTION:
The purpose of this study is to determine the maximal tolerated dose (MTD) of CIRT in the treatment of localized prostate cancer and to evaluate the efficacy of such treatment at the MTD. Participants will be treated with CIRT with escalating dose regimens to evaluate the maximal tolerated dose (MTD) in terms of acute and subacute toxicity observed during and within 6 months after the completion of CIRT. Once the MTD for localized prostate cancer is determined, the MTD will be used as the recommended dose to patients fulfilling the inclusion criteria in the Phase II part of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the prostate
* No lymph node and distant metastasis
* Age ≥ 20 and < 85 years of age
* Karnofsky Performance Score ≥70
* No previous pelvic radiation therapy (RT)
* No previous prostatectomy
* No previous invasive cancer (within 5 years before the prostate cancer diagnosis)except for skin non-melanoma cancer
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* No pathologically confirmed adenocarcinoma of the prostate
* Pelvic lymph node metastasis (N1)
* Distant metastasis (M1)
* Urinary obstructive symptoms (IPSS > 20)
* Previous pelvic radiotherapy
* Previous prostatectomy
* Severe systemic disorders
* Concomitant disorders including: chronic urinary or intestinal inflammatory conditions (for example, ulcerous recto-colitis, Crohn disease), anti-coagulant treatment (warfarin, heparin)
* Previous malignancy except for skin non-melanoma cancer or 3-year disease free interval from previous malignancy like non muscle invasive bladder cancer
* Non conformity of the radiotherapy dose distribution when compared to the dose constraints
* Psychiatric disorders or any other condition that can make unreliable the informed consent

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the date of CIRT to 6 months after the completion of CIRT, up to 6 months

SECONDARY OUTCOMES:
Overall survival of all patients | From the diagnosis of localized prostate, a median of 2 years
biochemical failure-free survival，bFFS | From the completion of CIRT, a median of 2 years
Progression-free survival of all patients | From the completion of CIRT, a median of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, Dr., Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Y, Li P, Yu Q, Wu S, Chen X, Zhang Q, Fu S. Preliminary exploration of clinical factors affecting acute toxicity and quality of life after carbon ion therapy for prostate cancer. Radiat Oncol. 2019 Jun 4;14(1):94. doi: 10.1186/s13014-019-1303-3. PMID 31164172